CLINICAL TRIAL: NCT05630521
Title: Testing Feasibility of the Medication Adherence Problem Solving for Hypertension (MASH) Intervention to Improve Antihypertensive Medication Adherence
Brief Title: Testing Feasibility of Medication Adherence Problem Solving for Hypertension
Acronym: MASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22031803
Record Dates: First submitted 2022-11-04; First posted 2022-11-29 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Adherence, Medication
Keywords: Medication adherence; Hypertension; Telehealth
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff will be blinded to the randomization sequence. Due to the nature of the intervention, participants and investigators delivering the intervention cannot be blinded.
  Study staff collecting outcome data will be blinded to participant group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Intervention Group (Experimental): The intervention components are: 1) educational modules and 2) bi-weekly telehealth visits for managed problem solving for 12 weeks.
  All intervention participants will be provided four educational modules, electronically and in print form. The modules are adapted from evidence-based materials developed by the American Heart Association, American College of Cardiology, and Centers for Disease Control and Prevention and cover (1) the causes of HTN, (2) how HTN raises risks for other chronic conditions, (3) medications for effectively managing high BP, and (4) how to manage barriers to medication adherence.
  Telehealth visits will supplement and reinforce the educational modules, addressing participants' specific knowledge needs and enhancing self-efficacy.
  Interventions: Behavioral: Medication Adherence Problem Solving for Hypertension
- Control (No Intervention): The study will use a usual-care control group. The standard of care for this patient population does not involve any type of medication adherence intervention or monitoring beyond regular clinic follow-up visits with their health care provider. Control group participants will be given printed handouts on the American Heart Association's Life's Simple 7 lifestyle changes for reducing cardiovascular risk, along with the instructions for using the MEMS cap. If control group participants ask about their antihypertensive medications during the study, they will be referred to their prescribing provider or pharmacist for any information that could not be obtained from the medication label or pharmacy packaging.

INTERVENTIONS:
Behavioral: Medication Adherence Problem Solving for Hypertension — The MASH program is a 12-week intervention containing two components: (1) four education modules on HTN causes, risks, treatment, and barriers to treatment; and (2) telehealth visits every 2 weeks with a registered nurse to deliver evidence-based managed problem solving strategies tailored on patients' responses to assessments of HTN beliefs, medication beliefs, and barriers impacting their medication adherence.
  Arms: Telehealth Intervention Group

SUMMARY:
Adherence to medications for high blood pressure is key to improving blood pressure control and reducing the impact of cardiovascular disease. This project will test the feasibility of a tailored telehealth intervention to help patients improve adherence to blood pressure medication.

DETAILED DESCRIPTION:
Improving rates of blood pressure (BP) control among adults with hypertension is a key step in reducing rates of myocardial infarction, stroke, and heart failure, and lowering overall mortality from cardiovascular disease. Unfortunately, over half of patients prescribed medication for hypertension do not take their medication as prescribed, leading to a high percentage of patients (45%) who are unable to reach their target BP despite being treated with antihypertensive medication. Low medication adherence has been linked with higher rates of myocardial infarction, stroke, and angina, as well as reduced life expectancy. Previously tested interventions to improve adherence to antihypertensive regimens have had limited efficacy, largely due to an underlying assumption that a single, standardized intervention approach will address all patients' reasons for nonadherence. Tailoring adherence interventions using a Managed Problem Solving approach will permit addressing each patient's reasons for nonadherence. This project will test the feasibility of the Medication Adherence Problem Solving for Hypertension (MASH) telehealth intervention, tailored to each participant's reasons for low adherence to their antihypertensive medication. The intervention is designed to assess beliefs about hypertension, beliefs about medications, and barriers to effective medication-taking We will then deliver intervention strategies to address each patient's problematic beliefs and barriers, applying the 5 steps of Managed Problem Solving. The proposed project aims are to 1) Assess the feasibility of MASH to improve antihypertensive medication adherence among adults with hypertension (HTN) by tracking recruitment, participant engagement and satisfaction with the intervention, as well as retention in the study; 2) Obtain estimates of efficacy of MASH compared to usual care on improving antihypertensive adherence as measured by electronic monitoring caps (MEMS) and lowering BP among persons with elevated BP at baseline over 12 weeks to inform future power analyses for a full-scale trial; and 3) Obtain estimates of other model parameters necessary to inform future power analyses for a full-scale intervention trial, including (a) intervention effects on targeted reasons for nonadherence (beliefs, barriers, perceived side-effects) and their subsequent association with medication adherence; (b) strength of covariate effects (e.g. education, household size, employment); and (c) the within-participant correlation between assessments. If successful, this intervention can also serve as a model for improving medication adherence in other chronic conditions and improve health outcomes for the half of patients with chronic conditions who struggle to manage their medications.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at time of study entry
2. Able to read, write, and converse in English
3. Have an active prescription for at least one HTN medication, reporting no antihypertensive prescription changes for 30 days prior to study entry
4. Have prescription drug coverage or participate in a prescription assistance program that covers medication costs.
5. Diagnosis of HTN, based on self-report or confirmed through medical records, where available. (Self-reported high BP has long been shown to be strongly correlated with presence of a HTN diagnosis.22-24 Self-report combined with presence of a prescribed HTN medication ensures that only participants with HTN will be included)
6. Must self-administer their own medications
7. Uncontrolled BP: systolic (SBP) ≥ 130 mmHg and/or diastolic (DBP) ≥ 80 mmHg at baseline
8. Nonadherent to HTN medication (Hill-Bone Medication Subscale score < 36) at screening

Exclusion Criteria:

1. Acutely ill (e.g., symptoms of myocardial infarction, respiratory distress, stroke)
2. Patients who have end-stage renal disease (ESRD) and/or are on dialysis
3. In state of hypertensive crisis (SBP >180 and/or DBP > 120 mmHg) at the time of study screening. Any participant in hypertensive crisis will be referred to their health care provider immediately for further instruction and follow-up, per current guidelines2
4. BP measurement is contraindicated on both upper extremities
5. Terminal chronic illness with a life expectancy of 6 months or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 12 weeks
  Number of patients enrolled in the study divided by number of patients invited to participate
Participant engagement | 12 weeks
  The number of intervention telehealth appointments kept divided by the number scheduled per-protocol
Patient satisfaction with intervention | 12 weeks
  Qualitative responses to questions about intervention delivery and content
Participant retention | 12 weeks
  % of randomized participants who complete the study

SECONDARY OUTCOMES:
Antihypertensive medication adherence | 12 weeks
  Adherence to antihypertensive medications as measured by electronic monitoring caps (MEMS)
Blood pressure | 12 weeks
  Resting blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Todd Ruppar, PhD, RN, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Final research data will be made available to other investigators who wish to conduct additional analyses. Coded data will be provided in the form of an Excel spreadsheet, and a codebook with explanations of the data fields. No individually-identifiable information will be included in the shared datasets. Data will be available for other investigators once any manuscripts using the requested data are accepted for publication. Requests for data will require a data-sharing agreement outlining the specific uses of the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for other investigators once any of the primary study investigators' manuscripts using the data are accepted for publication.
  Duration of availability to be determined.
Access Criteria: Requests for data will require a data-sharing agreement outlining the specific uses of the data.